CLINICAL TRIAL: NCT04269005
Title: SomPsyNet - Prevention of Psychosocial Distress Consequences in Somatic Medicine: a Model for Collaborative Care
Acronym: SomPsyNet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Gesundheitsförderung Schweiz, GFCH (Unknown); Bethesda Krankenhaus (Other); University Department of Geriatric Medicine FELIX PLATTER (Other); Gesundheitsdepartement Basel-Stadt (Unknown); Swiss Tropical & Public Health Institute (Other); Institute of Pharmaceutical Medicine (ECPM), University of Basel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019-01724; me19Schaefert
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psychosocial Distress
Keywords: mental health; mental disorder; mental comorbidity; mental-somatic multimorbidity; "stepped and collaborative care model" (SCCM)
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Hospital employees who will assign patients to the wards and clusters are blinded to randomization. Blinding of staff involved in the recruitment process is limited as phase 1 and phase 2 will consist of different study information and consent sheets. Trained staff will perform the follow-up assessment, and we intend to blind them regarding study phase allocation of the patients (if procedural aspects allow it).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): phase 0: Treatment as usual in combination with baseline and follow-up Survey but without any screening procedures (facilitating the study as a run-in phase to establish study procedures).
  phase 1: randomized and main control condition with TAU + collection of information on psychosocial distress in the baseline
  Intervention effects will be estimated, using the distressed focus sample, contrasting Phase 2 vs. Phase 1.
  We intend to conduct additional statistical analyses to compare data from phases 2 and 1 vs. phase 0 to estimate potential effects of introducing parts of the screening 1 without consequences.
- Intervention condition (Experimental): phase 2: implementation of the SCCM
  The intervention (SSCM) will be implemented step-wise in predefined sections at all three sites using a stepped-wedge cluster randomized trial design. Clusters will be randomized to different sequences that dictate the timing at which each cluster will switch from the control to the intervention condition.
  Interventions: Other: Implementation of the SCCM

INTERVENTIONS:
Other: Implementation of the SCCM — Implementation of the SCCM includes a baseline survey, assessment of screening questions stage 1 (with consequence), screening questions stage 2 (with consequence) and if necessary psychosomatic-psychiatric consultation and liaison service including if applicable post hospital intervention and a follow-up survey in a distressed focus sample.
  Arms: Intervention condition

SUMMARY:
This study is to evaluate the impact of the "stepped and collaborative care model" (SCCM) on health-related quality of life in somatic hospital patients with psychosocial distress.

DETAILED DESCRIPTION:
Given the burden of psychosocial distress, the public health relevance, and the current standard of health care, new approaches to a model of care for patients with mental-somatic multimorbidity are urgently needed. SomPsyNet is a comprehensive healthcare project for patients from somatic hospitals that promotes the prevention of psychosocial distress by establishing a stepped and collaborative care network in Basel-Stadt, Switzerland and may therefore help to counteract against the described lack of care.

SomPsyNet is a "stepped and collaborative care model" (SCCM) including a Psychosomatic-psychiatric consultation and liaison Service (CL Service) and post hospital intervention supported by a collaborative network structure. It aims to identify patients with psychosocial distress at an early stage during their hospital stay in a standardized way.

Implementation of the SCCM within this study using the stepped-wedge cluster randomized trial (SW-CRT) design will take place in phases:

* SomPsyNet phase 0: treatment as usual (TAU) in combination with the baseline and follow-up survey in a distressed focus sample.
* SomPsyNet phase 1: TAU in combination with the baseline survey, implementation of screening questions stage 1 ('baseline distress information from professionals', without consequence) in hospital routine and follow-up survey in a distressed focus sample.
* SomPsyNet phase 2 refers to the implementation of the SCCM: baseline survey, assessment of screening questions stage 1 (with consequence), screening questions stage 2 (with consequence) and if necessary psychosomatic-psychiatric consultation and liaison service including if applicable post hospital intervention and a follow-up survey in a distressed focus sample.

ELIGIBILITY:
Inclusion Criteria:

* patients from selected wards (i. e., somatic diseases treated at these wards from three somatic hospitals)

Exclusion Criteria:

* Inability to understand and speak German or any other language at which study is tailored at that point in time
* Inability to give informed consent by himself / herself
* Inability to follow the procedures of the study, e.g. due to severe medical / clinical limitations
* Need for immediate support as indicated by the risk of current suicidality or attempted suicide
* Oncological condition
* Already participated in the SomPsyNet project on the occasion of a previous hospitalization
* Confirmed current COVID-19 disease at time of screening for exclusion criteria
* Being hospitalized under the medical supervision of services of a ward that is not part of one of the SomPsyNet study clusters ('original ward'), but physically located in rooms of a ward contributing to one of the study clusters only because of lack of space in the original ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in health related quality of life | Baseline to 6 months follow-up
  Health related quality of life will be assessed with the 'Mental Health Component Summary score' of the Short Form-36 (SF-36). The SF-36 consists of 36-Items to measure health-related quality of life using eight concepts (physical functioning (PF, 10 items), physical role functioning (RP, 4 items), bodily pain (BP, 2 items), general health perception (GH, 5 items), vitality (VT, 4 items), social role functioning (SF, 2 items), emotional role functioning (RE, 3 items) and mental health (MH, 5 items) to measure the 'Mental Health Component Summary score'

SECONDARY OUTCOMES:
Change in Depression | Baseline to 6 months follow-up
  Current depressive disorders assessed by the eight-item Patient Health Questionnaire depression scale (PHQ-8)
Change in Generalized Anxiety Disorder | Baseline to 6 months follow-up
  Generalized Anxiety Disorder assessed by the 7-item Generalized Anxiety Disorder Scale (GAD-7)
Change in Somatic symptom disorder | Baseline to 6 months follow-up
  Psychological features of Somatic Symptom Disorder (SSD) assessed by the 12-item Somatic Symptom Disorder Scale (SSD-12)
Change in Somatic symptom burden | Baseline to 6 months follow-up
  Somatic symptom severity assessed by the 8-item Somatic Symptom Scale-8 (SSS-8)
Change in Quality of life | Baseline to 6 months follow-up
  "Health-related quality of life assessed by the 5-level EuroQol 5-dimensional questionnaire (EQ-5D- 5L)"
Change in health related quality of life | Baseline to 6 months follow-up
  Health-related quality of life assessed by the Physical Health Component Summary score of the SF-36
Health economics | 6 months to 3 years following initiation of the SCCM in a given patient
  total costs of hospital treatment including additional medical, psychiatric or physiotherapeutic treatment during patient's hospital stay; follow-up costs at treating hospitals; healthcare costs, relevant sub-categories of costs and medical resource use based on health insurance claims data; indirect costs due to reduced productivity
Resilience | 6 months follow-up
  Resilience assessed by the Resilience Scale for Adults (RSA)
Social support | 6 months follow-up
  Social support assessed by the Oslo social support scale (OSSS-3)

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Prof. Dr. rer. nat., Principal Investigator — Department of Psychosomatic Medicine, University Hospital Basel
Locations (4):
- Switzerland (4):
  - Universitäre Altersmedizin Felix Platter, Basel
  - Department of Psychosomatics/ Division of Medicine; University Hospital of Basel, Basel
  - Universitätsspital Basel - Frauenklinik, Basel
  - Bethesda Spital AG, Basel

IPD SHARING:
Plan to Share IPD: Yes
The datasets being held by the SomPsyNet project are not readily available. In the case of inquiries by third parties that wish to reuse data SomPsyNet data after an embargo period, the following procedure is planned. Researchers interested in the data may submit a project synopsis addressed to the publications committee of the SomPsyNet project and will have to obtain authorization from the responsible ethics committee as ordained in the Ordinance of 20 September 2013 on Human Research with the exception of Clinical Trials (Human Research Ordinance, HRO). The publication committee will review the project synopsis and will answer the formal requests of applicants.
Access Criteria: Only upon collection of all important consents and upon approval of the responsible ethics committee(s), the requested data will be transferred to the applicants. Third parties have to confirm and provide evidence to comply with all relevant Swiss and cantonal laws and regulations (especially regarding data protection and Human Research), as well as all obligations and regulations set out in the documents and contracts related to SomPsyNet. Fees may apply to cover expenses related to data reuse. Requests to access the datasets should be directed to Gunther Meinlschmidt, gunther.meinlschmidt@unibas.ch

REFERENCES:
- [Background] Aebi NJ, Caviezel S, Schaefert R, Meinlschmidt G, Schwenkglenks M, Fink G, Riedo L, Leyhe T, Wyss K; SomPsyNet Consortium. A qualitative study to investigate Swiss hospital personnel's perceived importance of and experiences with patient's mental-somatic multimorbidities. BMC Psychiatry. 2021 Jul 12;21(1):349. doi: 10.1186/s12888-021-03353-5. PMID 34253168
- [Background] Aebi NJ, Fink G, Wyss K, Schwenkglenks M, Baenteli I, Caviezel S, Studer A, Trost S, Tschudin S, Schaefert R, Meinlschmidt G; SomPsyNet Consortium. Association of Different Restriction Levels With COVID-19-Related Distress and Mental Health in Somatic Inpatients: A Secondary Analysis of Swiss General Hospital Data. Front Psychiatry. 2022 May 3;13:872116. doi: 10.3389/fpsyt.2022.872116. eCollection 2022. PMID 35592378
- [Derived] Meinlschmidt G, Frick A, Baenteli I, Karpf C, Studer A, Bachmann M, Dorner A, Tschudin S, Trost S, Wyss K, Fink G, Schwenkglenks M, Caviezel S, Rocco T, Schaefert R; SomPsyNet consortium. Prevention of psychosocial distress consequences in somatic hospital inpatients via a stepped and collaborative care model: protocol of SomPsyNet, a stepped wedge cluster randomised trial. BMJ Open. 2023 Nov 23;13(11):e076814. doi: 10.1136/bmjopen-2023-076814. PMID 37996236